CLINICAL TRIAL: NCT02861339
Title: Prevalence of Keratoconus in Inflammatory Bowel Diseases
Acronym: OSCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-A01680-45
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Inflammatory Bowel Diseases; Keratoconus
MeSH Terms: conditions — Inflammatory Bowel Diseases; Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Keratoconus and IBD (Experimental): Opthalmologic measure with DM OPD scan III (Nidek)
  Interventions: Device: Opthalmologic measure with DM OPD scan III (Nidek)

INTERVENTIONS:
Device: Opthalmologic measure with DM OPD scan III (Nidek) — Bilateral measure of corneal refractometry, pachymetry, topography and aberrometry

SUMMARY:
A retrospective study has shown the association between the inflammatory bowel diseases (IBD) and the presence of a keratoconus. This new study will measure the prevalence of keratoconus and follow its activity in patients affected by IBD and followed up in hepatology-gastroenterology department at Nancy Hospital. The prevalence of keratoconus will be compared to known data of literature about general population.

The secondary purpose is to search for a relationship between the presence of a keratoconus and activity criteria of IBD.

Perspectives are a systematic screening for keratoconus in patients affected by IBD with the amelioration of the ophthalmologic care of IBD patients and confirmation of the recent hypothesis of inflammatory origin of keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Affiliation to social security plan
* Diagnosis of IBD since more than 3 years, under treatment or not

Exclusion Criteria:

* Protected person
* Pregnant or breastfeeding women
* Person in life-and-death emergency
* Person deprived of liberty
* Refusal to remove contact lenses, where necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Absence or presence of keratoconus in IBD patients | day 0
  Data from OPD scan III corneal analyzer according to Rabinowitz and Klyce Maeda criteria. The presence of a keratoconus in at least one eye is considered positive.

SECONDARY OUTCOMES:
IBD clinical features using the Montreal classification for IBD | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Karine ANGIOI-DUPREZ, Principal Investigator — Service d'ophtalmologie- Hôpitaux de Brabois - CHU de NANCY

IPD SHARING:
Plan to Share IPD: No